CLINICAL TRIAL: NCT05860192
Title: Virtual Reality Mindfulness in Preoperative Anxious Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Regionale di Mendrisio (Other)
Responsible Party: Principal Investigator, Andrea Polito, Anesthesia Clinical Professor, Principal Investigator, Ospedale Regionale di Mendrisio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APolito1
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Test Anxiety; Anxiety State; Preoperative Period
MeSH Terms: conditions — Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality (Experimental): Each patient undergoes to a virtual reality session of mindfullness. This lasts about 30 minutes.
  Interventions: Device: Virtual Reality; Other: application for mindfulness

INTERVENTIONS:
Device: Virtual Reality — Use of this virtual reality headset to deliver a single mindfulness session
  Other Names: Meta, Oculus 2
Other: application for mindfulness — Application used to realize mindfulness in virtual reality
  Other Names: Guided Meditation VR

SUMMARY:
The goal of this interventional study is to reduce preoperative anxiety by Virtual Reality mindfulness.

Population: all adults, able to give their consent and scheduled for surgery with high preoperative anxiety defined by Amsterdam Preoperative Anxiety and Information Scale (APAIS) score > 10. The study will recruit 100 patients in one university teaching hospital.

The main question it aims to answer is: may mindfulness by Virtual Reality reduce preoperative anxiety in patients particularly anxious for the surgery? Participants will be asked to undergo to a single mindfulness virtual reality session before the surgery.

ELIGIBILITY:
Inclusion Criteria:

* adults able to give their consent, scheduled for elective surgery and with high preoperative anxiety defined by Amsterdam Preoperative Anxiety and Information Scale (APAIS) > 10

Exclusion Criteria:

* Pregnancy
* Epilepsy
* Pacemaker wearers
* Mental diseases
* Alcohol or drug addiction
* Severe hearing loss or blindness
* Simultaneous participation to other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change from one week before surgery in anxiety on STAI score some hours before the intervention | Up to two weeks
  The State-Trait Anxiety Inventory (STAI) score is a validated, self reported instrument to assessing state and trait anxiety. Possible scores range from "no or low anxiety" (20-37) to "high anxiety" (45-80). Change = (one week before - some hours before the surgery and after mindfulness in virtual reality)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Polito, Principal Investigator — Ospedale Beata Vergine
Locations (1):
- Andrea Polito, Mendrisio, Switzerland

IPD SHARING:
Plan to Share IPD: No